CLINICAL TRIAL: NCT02530502
Title: Phase I Trial of Radiation Therapy Plus Temozolomide With MK-3475 in Patients With Newly Diagnosed Glioblastoma (GBM)
Brief Title: Radiation Therapy With Temozolomide and Pembrolizumab in Treating Patients With Newly Diagnosed Glioblastoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The protocol was amendment to be stopped after phase I (phase 2 removed from protocol)
Sponsor: Northwestern University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Karan Dixit, Karan Dixit, MD, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 15C01; NCI-2015-00736 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STU00200883; NU 15C01 (Other: Northwestern University); P30CA060553 (NIH)
Record Dates: First submitted 2015-08-19; First posted 2015-08-21 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Adult Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — pembrolizumab; Radiotherapy; Radiation; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (RT, temozolomide, pembrolizumab) (Experimental): RT PORTION: Patients undergo focal RT over 42 days, and receive concurrent temozolomide PO QD on days 1-42 and pembrolizumab IV over 30 minutes on days 1, 22, and 43.
  POST-RT: After completion of RT, patients receive temozolomide PO QD on days 1-5 and 29-34 of course 1 and days 1-5 and 29-33 of subsequent courses, and pembrolizumab IV over 30 minutes on days 1, 22, and 43. Treatment repeats every 9 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity. After 6 courses, patients deriving benefit may continue to receive pembrolizumab for an additional 12 months.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab; Radiation: Radiation Therapy; Drug: Temozolomide

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Radiation: Radiation Therapy — Undergo focal RT
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; Irradiation; RADIATION; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Drug: Temozolomide — Given PO
  Other Names: CCRG-81045; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temodal; Temodar

SUMMARY:
The purpose of phase I trial is to determine the safest, most effective dose of MK-3475 (pembrolizumab), when used with radiotherapy and temozolomide for treating newly diagnosed patients with glioblastoma (GBM). Temozolomide binds to the deoxyribonucleic acid (DNA), changes it, and triggers the death of tumor cells. MK-3475 is an investigational drug, it is not currently approved by the Federal Drug Administration (FDA) for use in treating GBM but it is approved for treating melanoma. MK-3475 works by targets the local tumor immune-protection in solid tumors. It is hoped the addition of MK-3475 to the usual treatment for GBM will improve the current treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of radiation therapy (RT) + temozolomide (TMZ) + MK-3475 (pembrolizumab) followed by MK-3475 + TMZ x 6 cycles (1 cycle is 9 weeks), MK-3475 can continue for an additional 12 months.

SECONDARY OBJECTIVES:

Safety of MK-3475 in GBM.

TERTIARY OBJECTIVES:

I. To determine if there is a correlation of programmed cell death 1 (PD1) or programmed cell death 1 ligand 1 (PDL1) expression and T-cell infiltrate in pathology from first and, if applicable, second surgical specimens with outcome.

II. Assess changes in peripheral T-cell activation and tryptophan metabolites. III. Correlate o-6-methylguanine-deoxyribonucleic acid (DNA) methyltransferase (MGMT) status with outcome.

OUTLINE: This is a phase I, dose-escalation study of pembrolizumab, followed by a phase II study.

RT PORTION: Patients undergo focal RT over 42 days, and receive concurrent temozolomide orally (PO) once daily (QD) on days 1-42 and pembrolizumab IV over 30 minutes on days 1, 22, and 43.

POST-RT: After completion of RT, patients receive temozolomide PO QD on days 1-5 and 29-34 of course 1 and days 1-5 and 29-33 of subsequent courses, and pembrolizumab IV over 30 minutes on days 1, 22, and 43. Treatment repeats every 9 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity. After 6 courses, patients deriving benefit may continue to receive pembrolizumab for an additional 12 months.

After completion of study treatment, patients are followed up every 2-4 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed newly diagnosed glioblastoma; patients with an initial diagnosis of a lower-grade glioma are eligible if a subsequent biopsy was determined to be glioblastoma and they received no prior treatment
* No prior treatment with radiation or chemotherapy for their GBM
* No prior treatment with carmustine wafers
* Patients who have undergone recent surgery:

  * Must be a minimum of 14 days from surgery
  * Craniotomy or intracranial biopsy site must be adequately healed and free of drainage or cellulitis, and the underlying cranioplasty must appear intact at the time of registration
  * Magnetic resonance imaging (MRI) within 72 hours of surgery OR 4 weeks from surgery
* Karnofsky performance status >= 70%
* Stable or decreasing dose of corticosteroids within 5 days prior to treatment
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 7 days prior to receiving the first dose of study medication; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Patients need not have measurable or evaluable disease
* Absolute neutrophil count (ANC) > 1.5 x 10^9/L
* Platelet count > 100 x 10^9/L; or
* Hemoglobin (Hb) > 9.0 g/dL within 7 days prior to enrollment; note: the use of transfusion or other intervention to achieve Hb >= 9 g/dL is acceptable
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (except in patients diagnosed with Gilbert's disease)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]), alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x ULN
* Alkaline phosphatase (ALP) =< 2.5 x ULN
* Serum creatinine < 1.5 x ULN
* International normalized ratio (INR), prothrombin time (PT), or activated partial thromboplastin time (APTT) as follows: in the absence of therapeutic intent to anticoagulate the patient: INR < 1.5 or PT < 1.5 x ULN or aPTT < 1.5 x ULN; in the presence of therapeutic intent to anticoagulate the patient: INR or PT and aPTT within therapeutic limits (according to the medical standard in the institution) and the patient has been on a stable dose of anticoagulants for at least 2 weeks before registration
* Females of child-bearing potential (FOCBP) and males must agree to use two adequate contraception methods (give examples, e.g. hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 120 days following completion of therapy; should a female patient become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately

  * NOTE: A FOCBP is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

    * Has not undergone a hysterectomy or bilateral oophorectomy
    * Has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months)
* Patients must have the ability to understand and the willingness to sign a written informed consent prior to registration on study

Exclusion Criteria:

* Any prior treatment for the patients GBM
* Has a known diagnosis of immunodeficiency (human immunodeficiency virus [HIV] 1/2 antibodies) or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment excluding steroids; attempts should be made to have patient on lowest possible dose of steroids
* History of another malignancy in the previous 3 years, with a disease-free interval of < 3 years; exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy
* Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents; subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule; subjects that require intermittent use of bronchodilators or local steroid injections will not be excluded from the study; subjects with hypothyroidism stable on hormone replacement or Sjogren's syndrome will not be excluded from the study
* Has evidence of or a history of interstitial lung disease, non-infectious pneumonitis or pneumonitis
* Has an active infection requiring systemic antibiotics within 7 days of registration
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator; examples include

  * Hypertension (defined as 160/95) that is not controlled on medication
  * Ongoing or active infection requiring systemic treatment
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situations or substance abuse disorders that would limit compliance with study requirements
  * Any other illness or condition that the treating investigator feels would interfere with study compliance or would compromise the patient's safety or study endpoints
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways)
* Has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Has received a live vaccine within 30 days prior to the first dose of trial treatment
* Patients receiving any other investigational agents within 30 days prior to the first dose of trial treatment
* Patients who have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to MK-3475 are not eligible; known hypersensitivity to any excipients of MK-3475

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-09-30 (Actual); Primary Completion 2016-05-10 (Actual); Study Completion 2020-02-12 (Actual)

PRIMARY OUTCOMES:
The dose-limiting toxicity of Radiation Therapy With Temozolomide and Pembrolizumab will be evaluated | 9 weeks
  Any dose-limiting toxicity (DLT) experienced during the first cycle (9 weeks) of study treatment, will be determined. The Maximum Tolerated Dose (MTD) will constitute the RP2D

SECONDARY OUTCOMES:
Toxicity of Pembrolizumab | Up to 30 days after the last dose of study drug
  Adverse events will be described descriptively by giving frequencies of each event by type, severity, frequency, timing and attribution graded according to CTCAE version 4.0.

OTHER OUTCOMES:
Methylguanine-DNA methyltransferase (MGMT) status | Baseline
  Correlate MGMT status with outcome based on tumor tissue that will be analyzed
PDL1 expression in tumor | Baseline
  Tumor tissue will be analyzed to assess for PDL-1 levels
Peripheral T-cell activation | Up to 108 weeks (12 courses post-RT)
  Tumor tissue will be analyzed to collect peripheral markers of T-Cell activation
T-cell infiltrate in tumor | Baseline
  Tumor tissue will be analyzed to assess for T-cell infiltration
Tryptophan metabolites | Baseline
  Tumor tissue will be analyzed to collect peripheral markers of tryptophan metabolites

CONTACTS AND LOCATIONS:
Overall Officials: Karan Dixit, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States